CLINICAL TRIAL: NCT06950983
Title: Navigating Financial and Health-Related Social Needs in Adolescent and Young Adult Cancer Survivors (AYA-NAV): A Digital Intervention Pilot Study
Brief Title: Navigating Financial and Health-Related Social Needs in Adolescent and Young Adult Cancer Survivors (AYA-NAV)
Acronym: AYA-NAV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Melissa Beauchemin, Assistant Professor of Nursing, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AAAV3629; R21NR021310 (NIH)
Record Dates: First submitted 2025-03-05; First posted 2025-04-30 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Cancer in Adolescence
Keywords: Cancer; Adolescents; Young adults; Financial needs; Social needs
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Focus groups for aim 1. Parallel study model for aim 2 and 3
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AYA-NAV (Experimental): Stratified by age (15-25 years and 26-39 years). Participants will receive the following intervention components:
  1. A voucher to provide nominal support for immediate needs
  2. A standard resource sheet that has been co-developed with the social work team at CUIMC and lists available community resources for people living with cancer
  3. Direct support from the study team to set up their Findhelp.org account and to navigate through the available resources
  4. A 3-month check-in session with the study team by telephone, text message, or directly through findhelp.org
  5. A referral option to the Patient Advocate Foundation for individualized case management services
  6. If the participant reports educational/vocational needs, they will receive person-to-person vocational navigation and support consultation, which will provide referrals and navigation support to educational resources.
  The 6-month study survey will include implementation outcomes and optional interview.
  Interventions: Behavioral: AYA-NAV
- Enhanced Usual Care (No Intervention): Stratified by age (15-25 years and 26-39 years). Participants will receive information on Findhelp.org and a resource sheet. Follow-up surveys will be administered at 6 months.

INTERVENTIONS:
Behavioral: AYA-NAV — Support for AYA and vocational navigation sessions from clinical team
  Arms: AYA-NAV

SUMMARY:
Aim 1: Refine the HRSN navigation model to integrate a digital platform (Findhelp.org) to meet the needs of AYAs. The investigators will conduct iterative co-design sessions with AYAs and caregivers to understand their views on the existing Findhelp.org website and the likely need for other human-to-human and digital strategies to augment platform engagement (e.g., text reminders) and to address vocational needs.

Aim 2: Evaluate the feasibility and acceptability of the refined hybrid intervention that includes digital + person-to-person HRSN navigation.

Aim 3: Explore the preliminary impact of the refined hybrid intervention, compared to elevated usual care (a one-time referral to FindHelp.org alone), on reduction in financial distress (AYA and caregiver) and on AYA global health (i.e., mental, social, physical).

DETAILED DESCRIPTION:
Nearly 90,000 adolescent and young adults (AYA: defined by the National Cancer Institute [NCI] as age 15-39 years) are diagnosed with cancer annually in the United States (US), 85% of whom are expected to become long-term survivors. Compared to their peers, these survivors have an increased burden of chronic health conditions. AYAs also face devastating financial toxicity, defined as the negative personal financial impact of healthcare costs, resulting not only from the cost of care, but also from interrupted education, exclusion from the workforce, and developmental disruption in achieving or maintaining independence. In fact, AYA cancer survivors experience disproportionately higher rates of financial toxicity and unemployment, associated with poorer overall survival and bankruptcy, compared to older cancer survivors. Among AYA survivors, those with public insurance, who live in areas of high deprivation, and/or who are Black or Hispanic/Latino (hereafter Hispanic) have lower rates of 5- and 10-year survival, likely due in part to adverse social determinants of health (SDOH) and unmet health-related social needs (HRSN: financial strain, food insecurity, un/underinsurance, unstable housing, and suboptimal education).

The research team has studied financial toxicity and HRSN among Spanish- and English-preferring AYAs and their caregivers to develop participant-informed interventions to address unmet HRSN. This study is pilot testing a needs navigation model, adapted from an adult-directed model, among Spanish- and English-speaking AYAs who screen positive for high financial toxicity or unmet HRSN and are receiving care at Columbia University Irving Medical Center (CUIMC) in New York City. This model includes tailored needs navigation delivered over 6 months by a community organization that provides telephone-based case management to people facing life-limiting illness. Though AYA participants are initially interested in this AYA-HRSN navigation model (consent rates >85%), uptake and sustained engagement are rarely observed. During monthly check-ins with participants, investigators identified two gaps in the current model. First, AYAs do not perceive the model to be acceptable in addressing their needs because it is not accessible digitally. Findhelp.org is an established, digital network of local resources that can be leveraged to address this gap. Second, AYAs and caregivers request support to address educational and vocational needs, a resource not available through our community partner. Informed by these preliminary findings and given that AYAs are digital experts, the objective of this R21 proposal is to adapt the needs navigation model to a digital platform, while adding vocational navigation, to better engage AYAs and address their unmet HRSN. Using mixed methods, the investigators will refine the intervention (Aim 1) and conduct a randomized pilot study to measure its feasibility and acceptability (Aim 2) and compare the impact of the digital HRSN navigation intervention with elevated usual care (Aim 3). This study will enroll and randomize (1:1) 80 English- and Spanish-speaking AYAs who are within 6 months of completing curative-intent cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

Aim 1:

* AYAs (age 18-39) who have/had a diagnosis of cancer are eligible to participate.
* English or Spanish-speaking

Aim 2 and 3:

* AYAs (age 15-39) who were diagnosed with cancer or began treatment for cancer within the past 6 months, or those who are still on first treatment for cancer (non-relapse)
* English or Spanish-speaking
* For AYAs who are < 18 years, caregiver participation will be required; for AYAs > 18 years, caregivers may co-participate if desired; the primary unit of focus is the AYA patient.

Exclusion Criteria:

* Dyad with caregiver or younger AYA that previously participated in study AAAU2405 or AAAY9477
* Unable to complete financial survey questions or contraindicated (as outlined in Protection of Human Subjects)
* Dyad with younger AYAs who are enrolled on hospice or receiving other end-of-life care

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-07-23 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate (feasibility) | Up to 6 months
  Percent eligible out of total screened
Consent rate (feasibility) | Up to 6 months
  Percent consented out of eligible total
Retention rates (feasibility) | Up to 6 months
  Percent of enrolled that completed the 6-month assessment
Comprehensive Score of Financial Toxicity (COST) score | baseline, 6-months
  The COST is a patient-reported outcome measure that describes the financial distress experienced by cancer patients. It is a 11-item questionnaire with a score range of 0-44. Lower COST values indicate higher toxicity. Higher scores indicate lower financial toxicity.

SECONDARY OUTCOMES:
Patterns of engagement | Up to 6 months
  Engaged with an intervention component at least once
Implementation outcomes | 6 months
  12-item AIM/IAM/FIM (Acceptability of Intervention Measure; Intervention Appropriateness Measure; Feasibility of Intervention Measure). Each item gets a score of 1-5. A higher score indicates greater acceptability, appropriateness, or feasibility.
Patient-Reported Outcomes Measurement Information System (PROMIS) Global Mental Health Measure | Baseline, 6-months
  PROMIS Global Health measure. Quality of Life Measure (scale 1-5; higher number indicating better QoL)

OTHER OUTCOMES:
Connor Davidson Resilience Scale (CD-RISC) | Baseline, 6-months
  Resiliency measure. Total score ranges 0-40. Higher score indicates higher resiliency.
Patient-Reported Outcomes Measurement Information System (PROMIS) Global Physical Health | Baseline, 6-months
  PROMIS Global Health measure. Quality of Life Measure (Scale 1-5; higher number indicates better quality of life;

CONTACTS AND LOCATIONS:
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No